CLINICAL TRIAL: NCT01516411
Title: Promoting Healthy Lifestyles Using Mobile Phones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Abby C King, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-09162011-8409
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Health Behavior
Keywords: Health Promotion; Physical Activity; Sedentary Time; Smartphones
MeSH Terms: conditions — Health Behavior; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cognitive app (Active Comparator): Cognitive app promotes behavior change via goal setting, feedback, and problem solving
  Interventions: Behavioral: Mobile Intervention for Lifestyle Eating/Exercise @ Stanford
- Social app (Active Comparator): Social app promotes behavior change via social relationships and feedback
  Interventions: Behavioral: Mobile Intervention for Lifestyle Eating/Exercise @ Stanford
- Affect app (Active Comparator): Affect app promotes behavior change via game-like elements including the use of a bird avatar as a visual representation of one's activities and operant conditioning
  Interventions: Behavioral: Mobile Intervention for Lifestyle Eating/Exercise @ Stanford
- Nutrition app (Active Comparator): Nutrition app promotes behavior change bvia tracking of food consumption
  Interventions: Behavioral: Mobile Intervention for Lifestyle Eating/Exercise @ Stanford

INTERVENTIONS:
Behavioral: Mobile Intervention for Lifestyle Eating/Exercise @ Stanford — Participants are randomized to one of 4 groups, each of which uses a different Smartphone app to promote health behavior change

SUMMARY:
The purpose of this research is to test programs to increase physical activity and reduce sedentary behavior using motivational messages over a cell phone.

DETAILED DESCRIPTION:
We want to learn if conceptually-based behavioral interventions for promoting increased physical activity and decreased sedentary behavior via state-of-the-art mobile phones will be efficacious at improving these behaviors relative to commercially available Android applications as a control. If efficacious, these types of intervention programs could be disseminated to a wide variety of sedentary and underactive adults at a relatively low cost. This could have a potentially significant impact on promoting improved health such as reduced obesity, a key problem within the U.S.

ELIGIBILITY:
Inclusion Criteria:

* aged 45 and older, currently sedentary, owns and uses a cell phone but not a Smartphone, willing to be randomly assigned

Exclusion Criteria:

* free of clinically evident cardiovascular disease or any other medical condition or disorder that would limit participation in moderate intensity physical activities akin to brisk walking

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time spent being physically active | 2 months
Time spent sitting | 2 months
Changes in food consumption | 2 months

SECONDARY OUTCOMES:
Beliefs and behaviors about Smartphones | 2 months
Beliefs and behaviors about the Smartphone application | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Abby C King, PhD, Principal Investigator — Stanford Prevention Research Center
Locations (1):
- Stanford Prevention Research Center, Palo Alto, California, United States

REFERENCES:
- [Derived] King AC, Hekler EB, Grieco LA, Winter SJ, Sheats JL, Buman MP, Banerjee B, Robinson TN, Cirimele J. Effects of Three Motivationally Targeted Mobile Device Applications on Initial Physical Activity and Sedentary Behavior Change in Midlife and Older Adults: A Randomized Trial. PLoS One. 2016 Jun 28;11(6):e0156370. doi: 10.1371/journal.pone.0156370. eCollection 2016. PMID 27352250